CLINICAL TRIAL: NCT04386655
Title: Telemedicine Brain Injury Coping Skills (BICS-T) Support Group for Brain Injury Survivors and Caregivers
Brief Title: Brain Injury Coping Skills - Telemedicine: Phase II
Acronym: BICS-T-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Devan Parrott (Other)
Responsible Party: Sponsor-Investigator, Devan Parrott, Director and Biostatistician, Rehabilitation Hospital of Indiana
Organization: Rehabilitation Hospital of Indiana (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1902473107
Record Dates: First submitted 2019-08-08; First posted 2020-05-13 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury; Coping Skills; Caregivers
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial Approximately 50 survivors with brain injury who meet inclusion/exclusion criteria and their caregivers will be recruited. There will be 3 waves within one year. Each wave will be split into 2 groups. Half of the participants in each wave will attend a regular BICS program (in-person), while the other half will participate in a BICS-T program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Group (Experimental): BICS-T is the intervention that will take place over telemedicine software on the iPad provided to participants
  Interventions: Behavioral: Brain Injur Coping Skills - Telemedicine
- In-Person Group (Active Comparator): Participants a part of the in-person BICS group will then come to the NRC for the following BICS sessions. This group is the traditional, in-person, BICS group
  Interventions: Behavioral: Brain Injur Coping Skills - Telemedicine

INTERVENTIONS:
Behavioral: Brain Injur Coping Skills - Telemedicine — BICS sessions (both in-person and telemedicine) will occur once a week for 12 weeks. Each session will last two hours.
  Modules of BICS include: Introduction to Brain Injury, Expectations for Recovery, Tips on Managing Challenging Problems, Learning about Depression after the Brain Injury, The 4 R's of Stress Management, Communicating Effectively with Professionals

SUMMARY:
For phase II, the objective is to compare the effectiveness of BICS-T with the well-established BICS in-person group. Information gained from phase I (the feasibility study) was used to make necessary changes to the BICS-T protocol.

The purpose of this study is to provide survivors of brain injury and caregivers greater support and teach adaptive coping strategies, through a designed and studied a coping skills group specifically for brain injury survivors and their caregivers at the Rehabilitation Hospital of Indiana (RHI) called the Brain Injury Coping Skills group (BICS).

DETAILED DESCRIPTION:
Brain injury can be devastating for both patients and family members and can result in chronic difficulties in vocational, social, financial, as well as physical functioning. The occurrence of emotional and neurobehavioral challenges in individuals with brain injury is also common with research consistently showing links between these challenges and a person's overall rehabilitation outcome. Additionally, family functioning and caregiver well-being has been shown to influence rehabilitation outcome for a survivor after brain injury. In fact, individuals with families and caregivers who receive support and services, as well as learn adaptive coping strategies, are less likely to exhibit these marked levels of psychological distress.

In order to provide patients and caregivers greater support and teach adaptive coping strategies, the authors of this grant designed and studied a coping skills group specifically for brain injury survivors and their caregivers at the Rehabilitation Hospital of Indiana (RHI) called the Brain Injury Coping Skills group (BICS). BICS is a 12 session (one session per week), manualized, cognitive-behavioral treatment group designed to provide support, coping skills, and psychoeducation aimed to improve perceived self-efficacy (PSE) and emotional functioning. Perceived self-efficacy is the belief or confidence in one's ability to deal with the challenges related to a specific situation (e.g., brain injury). PSE has been found to be strongly linked to social participation, increased positive regard toward the caregiving role, and was found to be the greatest contributing factor to predicting life satisfaction. Cicerone and Azulay found that the greatest contribution to predicting life satisfaction was the person's PSE for managing their cognitive challenges.

Telemedicine is one possible option for rural patients. With increases in the availability of internet and electronic communication, patients now have immediate access to experts and treatment providers who specialize in brain injury. In fact, results from a needs assessment from Ricker and colleagues in 2002 identified telemedicine as a desired need of the brain injury community. To date, several studies have used telemedicine as an avenue to address brain injury rehabilitation for rural patients and caregivers.

For phase II, the objective is to compare the effectiveness of BICS-T with the well-established BICS in-person group. Information gained from phase I (the feasibility study) was used to make necessary changes to the BICS-T protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participants enrolled in the study will be (1) persons with a history of brain injury (e.g., Traumatic Brain Injury; TBI) or acquired BI (e.g., stroke, hypoxia, ruptured aneurysm, or metabolic encephalopathy) OR a caregiver of a brain injury survivor; (2) 18 years of age and older; and (3) at least six months post-injury. Since there is no reason to believe that treatment effectiveness varies with chronicity, no maximum has been set for time post-injury.

Exclusion Criteria:

* Participants will not be included in the study if they present with the following: (1) at imminent risk of psychiatric breakdown, or in imminent danger of hurting themselves or others; (2) active psychosis; (3) aphasia that limits group participation; or (4) significant neurobehavioral difficulties that would be deemed disruptive to group participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Brain Injury Self-Efficacy Scale (BICS-Q) | Through study completion, up to 5 months
  This measure assesses perceived self-efficacy regarding a person's brain injury. Participants respond to each item using a scale from 0 (Not at all) to 4 (Extremely). Items are totaled and higher scores suggest greater perceived self-efficacy.

SECONDARY OUTCOMES:
The Group Climate Questionnaire (GCQ) | 3 months
  the most commonly used group process instrument. It is a self-report, 12-item questionnaire that assesses the person's perceptions of the group's therapeutic environment. Items are scored on a 7-point Likert scale ranging from "Not at all" to "Extremely." The three subscales includes Engagement (the level of positive working group atmosphere), Conflict (the level of anger and tension in the group), and Avoidance (the level of behaviors indicating avoidance of personal responsibility of group work by the members).
Group Session Rating Scale (GSRS) | 3 months
  This is a 4-item questionnaire that assesses a person's feelings and perceptions towards the group content and relationships. Items are measured on an analog scale, ranging from 1-10. The four items measure four different aspects of the group environment including: Relationship, Goals, Acceptability, and Overall Fit.
Patient-reported outcome measurement information system (PROMIS): General Self-Efficacy | Through study completion, up to 5 months
  This measures a person's confidence in managing daily activities, emotions, medications/treatments, social interactions, and symptoms. Participants respond to each item using a scale from 1 (I am not at all confident) to 5 (I am very confident). Higher scores suggest higher perceived self-efficacy.
Quality of Life After Brain Injury (TBIQOL) | Through study completion, up to 5 months
  This is a quality of life measure designed specifically for patients with brain injury. Participants respond to how satisfied they feel about each item using the following scale: 1 (Not at all), 2 (Slightly), 3 (Moderately), 4 (Quite), 5 (Very). Item scores are added and higher scores suggest higher perceived quality of life after brain injury.
Patient-reported outcome measurement information system (PROMIS): Health-Related Quality of Life (HRQL) Physical Function | Through study completion, up to 5 months
  This is a part of an evaluation on a person's overall quality of life based on physical limitations and ability to participate socially. Participants rate each statement from 1 (unable to do) to 5 (without any difficulty). Higher scores suggest greater physical functioning ability.
Patient-reported outcome measurement information system (PROMIS): Health-Related Quality of Life (HRQL) Anxiety scale | Through study completion, up to 5 months
  This is a part of an evaluation on a person's overall quality of life based on physical limitations and ability to participate socially. Participants rate each statement from 1 (Never) to 5 (Always). Higher scores suggest greater anxiety.
Patient-reported outcome measurement information system (PROMIS): Health-Related Quality of Life (HRQL) Depression scale | Through study completion, up to 5 months
  This is a part of an evaluation on a person's overall quality of life based on physical limitations and ability to participate socially. Participants rate each statement from 1 (Never) to 5 (Always). Higher scores suggest greater depressive symptoms.
Patient-reported outcome measurement information system (PROMIS): Health-Related Quality of Life (HRQL) Fatigue scale | Through study completion, up to 5 months
  This is a part of an evaluation on a person's overall quality of life based on physical limitations and ability to participate socially. Participants rate each statement from 1 (Not at all) to 5 (Very much). Higher scores suggest greater fatigue.
Patient-reported outcome measurement information system (PROMIS): Health-Related Quality of Life (HRQL) Sleep Disturbance scale | Through study completion, up to 5 months
  This is a part of an evaluation on a person's overall quality of life based on physical limitations and ability to participate socially. Participants rate each statement from 1 (Not at all) to 5 (Very much). Higher scores suggest greater sleep disturbance (worse sleep).
Patient-reported outcome measurement information system (PROMIS): Health-Related Quality of Life (HRQL) Ability to Participate in Social Roles and Activities scale | Through study completion, up to 5 months
  This is a part of an evaluation on a person's overall quality of life based on physical limitations and ability to participate socially. Participants rate each statement from 1 (Always) to 5 (Never). Higher scores suggest greater ability to participate in social roles and activities.
Patient-reported outcome measurement information system (PROMIS): Health-Related Quality of Life (HRQL) Pain Interference scale | Through study completion, up to 5 months
  This is a part of an evaluation on a person's overall quality of life based on physical limitations and ability to participate socially. Participants rate each statement from 1 (Not at all) to 5 (Very much). Higher scores suggest greater likelihood that pain is interfering with the participant's every functioning.
Patient-reported outcome measurement information system (PROMIS): Health-Related Quality of Life (HRQL) Pain Intensity scale | Through study completion, up to 5 months
  This is a part of an evaluation on a person's overall quality of life based on physical limitations and ability to participate socially. Participants rate their pain on a 0 to 10 scale (0 = no pain, 10 = worse pain imaginable).
Therapeutic Factors Inventory (TFI) | 3 months
  This a 7-point Likert scale for group settings. It measures one's feeling of acceptance in a group setting, as well as sense of belonging, working together, trust, and caring. The scale ranges from 1 (Strongly Disagree) to 7 (Strongly Agree). Higher scores suggest greater positivity about group acceptance, trust, caring, and working together.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No